CLINICAL TRIAL: NCT04608383
Title: Laparoscopy and COVID-19 Contamination
Acronym: LAPCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200611
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: LAPAROSCOPY; pneumoperitoneum
MeSH Terms: conditions — COVID-19; Pneumoperitoneum | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess peritoneal fluid, usually taken during laparoscopy Exsufflation of the pneumoperitoneum through a filter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Additional and minimal collection of products of the human body carried out during a sample for standard of care — * Swab of the peritoneal fluid for traces of COVID19. The collection of peritoneal fluid is a standard care practice.
  * Swab from the laparoscopy filter

SUMMARY:
The aim of the study is to search the presence of the SARS-COV-2 virus (COVID19) in the pneumoperitoneum of patients with a positive (or suspected) COVID19 status during a routine laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age
* Indication for laparoscopy
* Positive (past or current) or suspected Covid19 status (cough, fever, suggestive radiological images, etc.)
* Lack of opposition to participating in the study

Exclusion Criteria:

* Patient under legal protection
* Covid19 status negative, (former or current) and not suspected
* Patient unable to object
* Patient with no social security care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult requiring a laparoscopic procedure with a positive or suspected Covid19 status.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The main objective of the study is to demonstrate the presence of SARS-COV-2 in the exsufflated gas at the end of laparoscopy. | Day 1 , at the end of the surgery
  The SARS-COV-2 will be looked for in the gas before its elimination at the end of the intervention. To this end, the PCR search will be carried out on the filter used

SECONDARY OUTCOMES:
The secondary objective of the study is to demonstrate the presence of SARS-COV-2 in the peritoneal fluid during laparoscopy | Day 1 , at the end of the surgery
  SARS-COV-2 will be tested for by PCR in the peritoneal fluid collected during laparoscopy

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - AP-HP, Bicêtre Hospital, Anesthesia Department, Le Kremlin-Bicêtre
  - AP-HP, Bicêtre Hospital, Department of Digestive and Oncological Surgery, Le Kremlin-Bicêtre
  - AP-HP, Bicêtre Hospital, Gynecology department, Le Kremlin-Bicêtre
  - AP-HP, Bicêtre Hospital, Urology Department, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No